CLINICAL TRIAL: NCT01558700
Title: Brain Morphometries in OA Patients Treated With Duloxetine
Brief Title: Duloxetine in Osteoarthritis (OA) Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU00039556
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; pain; brain; gray matter
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine capsule 30mg once a day for one week, then 60mg once a day for 15 weeks, then 30mg once a day for one week.
  Interventions: Drug: Duloxetine
- Sugar pill (Placebo Comparator): Matching capsule given once a day for a total of 17 weeks.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Duloxetine — Duloxetine capsule 30mg once a day for one week, then 60mg once a day for 15 weeks, then 30mg once a day for one week.
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Sugar pill — Matching capsule given once a day for a total of 17 weeks.
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
This study aims to determine in people with knee Osteoarthritis (OA) if relief of pain after treatment with either duloxetine or placebo is associated with changes in brain anatomy.

DETAILED DESCRIPTION:
This study and the hypotheses to be tested arise from work done in our group evaluating brain cortical changes in people with chronic back pain. These studies demonstrated a loss of about 1.5 cc of neocortical gray matter per year of living with the condition, not including gray matter lost due to aging. Since this original publication, more than ten studies have replicated this basic result, showing that distinct chronic pain conditions are associated with specific brain anatomical reorganization, characterized by regional decreases in grey matter density. Recently, other studies have shown that when chronic pain is completely reversed, these anatomical changes seem to at least partially reverse within the time span of 4-12 months, providing evidence for a time window for reversal of grey matter abnormalities A fundamental question that arises from these recent studies is the extent of reversibility of the brain atrophy associated with chronic pain following continuous use of a pain-relieving drug. Apkarian's lab has generated strong evidence that the brain anatomy of subjects with osteoarthritis (OA) is dramatically different from that of healthy subjects. Given that recent data show that hip replacement OA reverses brain atrophy, the investigators can now hypothesize with greater confidence that an effective analgesic should also reverse at least some of the brain atrophy observed in OA. Thus, a study in patients with chronic knee OA treated with duloxetine provides a unique opportunity to answer this question. Since OA patients in this study will have a single new agent for four months, one can directly examine the effects of treatment in relation to progression or regression of brain atrophy. One can also examine whether or not a placebo, which is thought to reflect attentional and motivational states, affects changes in atrophy, and if so, to what extent.

The investigators consider the brain atrophy in chronic pain to be an overall marker of the extent of nervous system reorganization a subject has developed while living with the condition. Animal models of various chronic pain conditions repeatedly provide evidence for this idea, showing, for example, dramatic changes in the way pain is processed in the periphery, the spinal cord, and at the level of individual neurons. The investigators presume that these changes are the same ones contributing to atrophy in human chronic pain. However, most of underlying mechanisms remain to be uncovered. In addition, humans suffering from chronic pain exhibit a large number of cognitive and emotional deficits. The investigators presume that these deficits are directly related to the brain atrophies discovered in chronic pain conditions. Unfortunately, there are no direct studies linking brain regional atrophies to cognitive abilities in chronic pain, although such preliminary studies are underway in Apkarian's lab. Thus, in addition to the answering the previous questions, the present study will also allow us to investigate the extent to which reversing atrophy corresponds to reversing plasticity at multiple levels in the nervous system, as well as whether such reversal also corresponds to improvements in cognitive and emotional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-80 years
* ACR criteria for OA including Kellgren-Lawrence radiographic OA grades II-IV
* VAS pain score >5/10 within 48 hrs of the phone screen and visit 1 (Screening)
* Knee OA for a minimum of 12 months
* Need for daily pain medication to manage symptoms of OA

Exclusion Criteria:

Currently taking MAO inhibitors or any centrally acting drug for analgesia, depression

* Narrow angle glaucoma
* Uncontrolled hypertension
* Co-existing inflammatory arthritis, fibromyalgia or other chronic pain state.
* If a female, pregnant, trying to become pregnant, or lactating
* Major depressive disorder
* Substantial alcohol use or history of significant liver disease
* Use of MAO inhibitors, triptans, serotonin precursors (tryptophan)
* Use of potent CYP1A2 inhibitors, Thioridazine, and anti-depressants
* Diabetes, type 1 or type 2
* Condition in which the Investigator believes would interfere with the subject's ability to comply with study instructions, or might confound the interpretation of the study results or put the subject at undue risk
* MRI safety necessitates the exclusion of subjects having one or more of the following:

  * Metal fragments in the eye or face, or having worked previously in the metal industry
  * Implantation of any electronic devices such as (but not limited to) cardiac pacemakers, cardiac, defibrillators, and cochlear implants or nerve stimulators.
  * Surgery on the blood vessels of the brain
  * Claustrophobia (fear of enclosed places)
  * Piercings or tattoos
  * More than 250 lbs in weight
  * Obvious brain abnormalities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schnitzer, MD, PhD, Study Director — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Leaney AA, Lyttle JR, Segan J, Urquhart DM, Cicuttini FM, Chou L, Wluka AE. Antidepressants for hip and knee osteoarthritis. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012157. doi: 10.1002/14651858.CD012157.pub2. PMID 36269595
- [Derived] Tetreault P, Mansour A, Vachon-Presseau E, Schnitzer TJ, Apkarian AV, Baliki MN. Brain Connectivity Predicts Placebo Response across Chronic Pain Clinical Trials. PLoS Biol. 2016 Oct 27;14(10):e1002570. doi: 10.1371/journal.pbio.1002570. eCollection 2016 Oct. PMID 27788130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Sugar Pill
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Sugar Pill | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (4.2) | 58.9 (8.6) | 58.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Gray Matter Volume
Description: The change in gray matter volume is evaluated by subtracting the volume after the treatment (week 16) to the volume before treatment (baseline)
Time Frame: 16 weeks compared to baseline
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Duloxetine | Sugar Pill
Number analyzed (Participants) | 19 | 21
percentage of change | -0.34 (0.21) | -0.92 (0.19)

2. Secondary Outcome: Change in Pain Magnitude
Description: The Western Ontario and McMaster Osteoarthritis Index (WOMAC) score change was assess by subtracting WOMAC score after treatment (week 16) to the baseline WOMAC score. WOMAC score has a range from 0 up to 96, higher score meaning worse condition. The outcome is the decrease in WOMAC scores, meaning that the higher is the decrease, the most improvement in the condition.
Time Frame: 16 weeks compared to baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine | Sugar Pill
Number analyzed (Participants) | 19 | 21
Scores on a scale | 8.3 (6.1) | 8.7 (6.4)

ADVERSE EVENTS:
Arm/Group | Duloxetine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 6/19 | 6/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=19) | Sugar Pill (N=21)
dizziness, groggy (Nervous system disorders) | 4 (4) | 3 (3)
worsening knee pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No